CLINICAL TRIAL: NCT05085340
Title: MULTIple Doses of IPTi Proposal: a Lifesaving High Yield Intervention
Acronym: MULTIPLY
Status: Completed | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Centro de Investigação em Saúde de Manhiça (Other); Medicines for Malaria Venture (Other); University of Lomé (UL), Togo (Unknown); University of Sierra Leone (Other)
Responsible Party: Sponsor
Other Study IDs: RIA2020S 3272
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Malaria
Keywords: IPTi; Sulfadoxine-pyrimethamine; IPTi-SP; chemoprevention; Intermittent preventive treatment of malaria in infants; children; EPI; Expanded Programme of Immunization; SSA; sub-Saharan Africa; infants; malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Intermittent preventive treatment of malaria in infants (IPTi) with sulfadoxine-pyrimethamine (SP) — IPTi will be administered as full therapeutic courses of SP alongside routine EPI immunisations at defined intervals corresponding to vaccination schedules - usually at 10 weeks, 14 weeks, and 9 months of age - to infants living in project districts. Additional doses of IPTi will be administered at 6, 12, and 15 or 18 months of age, coinciding with vitamin A administration and measles booster immunisation. The number of doses of IPTi a child will receive will depend of the EPI schedule in the country, with a maximum of six doses in the first two years of life.
  Other Names: IPTi-SP

SUMMARY:
As efforts to control malaria are stalling, and the disease is particularly severe in children under the age of two, it is imperative for countries in sub-Saharan Africa, with areas of moderate-to-high transmissions, to implement Perennial Malaria Chemoprevention (PMC) delivered through the Expanded Program on Immunization (EPI), which is the only feasible, sustainable and cost-effective strategy to reach this high-risk group. PMC is a full therapeutic course of antimalarial medicine (with sulfadoxine-pyrimethamine, SP) delivered to infants in the context of routine immunisation services during the first two year of life.

PMC has been shown to be safe, efficacious in reducing clinical malaria, anaemia and hospital admissions, and to be highly cost-effective; for all these reasons, the World Health Organization (WHO) recommended in 2010 Intermittent Preventive Treatment for Infants (IPTi) for malaria prevention. Only one African country - Sierra Leone -put IPTi into policy and practice. Concerned with this slow adoption, WHO in 2019 recommended adaptations be urgently tested through pilots assessing impact, operational feasibility and cost effectiveness. In 2022, WHO expanded that recommendation to cover children through the age of two because of studies documenting the value in children aged 12 to 24 months. The name for this preventive treatment has consequently changed to Perennial Malaria Chemoprevention (PMC) as the updated recommendation is no longer just for infants.

MULTIPLY is the pilot implementation of PMC in selected districts in Mozambique, Sierra Leone and Togo to maximise the delivery and uptake of PMC, to achieve the full potential of this intervention. Working with the ministries of health in Mozambique, Sierra Leone and Togo, MULTIPLY will give up to 6 doses of PMC in the first two years of life. PMC will be given at health facilities and EPI mobile outreach clinics using a paediatric dispersible formulation of SP, alongside routine vaccinations and vitamin A supplementation.

DETAILED DESCRIPTION:
The study will be conducted in 3 sub-Saharan African countries; Sierra Leone, Mozambique and Togo.

Sample size; Assuming an average population of a district/project area of 150,000 inhabitants and a percentage of U2 children of 5%, the project intervention will target approximately 45,000 U2 children in total (i.e. 7,500 children per country and per year for 2 years).

Study population; Children U2 who are eligible for IPTi in the selected MULTIPLY district of each country.

ELIGIBILITY:
Inclusion Criteria:

All infants attending their 2nd EPI contact who are eligible to receive the corresponding immunisations.

Exclusion Criteria:

Infants/children; with acute malaria; known to have sulfa allergies; who have taken SP in the past 4 weeks; who are HIV-exposed or HIV-infected

Ages: 10 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants attending their 2nd EPI contact who are eligible to receive the corresponding immunisations.
Sampling Method: Probability Sample
Enrollment: 94252 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of children having received at least three doses of IPTi | Month 24

SECONDARY OUTCOMES:
Malaria prevalence in under 2 year old children living in project districts | Month 24
Malaria incidence in under 2 year old children living in project districts | Month 24
Coverage of EPI routine vaccines in children living in project districts | Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menéndez, MD, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (3):
- Fundaçao Manhiça, Manhiça, Manhiça, Mozambique
- College of Medicine & Allied Health Sciences (COMAHS), University of Sierra Leone, Freetown, Sierra Leone
- University of Lomé, Lomé, Togo

IPD SHARING:
Plan to Share IPD: No